CLINICAL TRIAL: NCT00113542
Title: An Open Label Study of Tetrathiomolybdate in the Treatment of Psoriasis Vulgaris
Brief Title: A Study of Tetrathiomolybdate in the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 508
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2008-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Tetrathiomolybdate
MeSH Terms: conditions — Psoriasis | interventions — tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate (TM)

SUMMARY:
Psoriasis is a common skin disease affecting an estimated 2.6% of the US population. It is a chronic, recurrent condition for which there is no cure, but there are ways to control it. Psoriasis is characterized by epidermal hyperplasia (abnormal increase in the number of normal cells of the outer layer of the skin). Tetrathiomolybdate (TM), a copper chelator (a drug that removes copper from the bloodstream) was first created to treat Wilson's disease, a disorder caused by too much copper in the blood. Studies in animals have since shown that TM may also prevent the formation of new blood vessels and may also block the key components of inflammation (swelling, redness, and pain) caused by psoriasis. TM is not approved by the FDA for any use yet. It is an investigational drug used for clinical research. We propose to test whether a new treatment with TM can in fact improve or stabilize psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of Tetrathiomolybdate in psoriasis therapy. Psoriasis is a common skin disease affecting an estimated 2.6% of the US population. It is a chronic, recurrent condition for which there is no cure but ways to control it. Psoriasis is characterized by epidermal hyperplasia, increased dermal angiogenesis, and infiltration of activated lymphocytes. Beginning with the observation that cyclosporin A, whose primary action is to inhibit lymphokine release and proliferation of T cells, was effective in the treatment of psoriasis, the last two decades saw a major paradigm shift in the pathogenesis of psoriasis, from a view of psoriasis as a disease of epidermal origin to a view of it as an epidermal response to immunological injury. In fully activated T cells in psoriatic skin, the T1/T2 cytokine balance is shifted in favor of T1 expression, with production of IL-2 and IFN-γ. Activated T1 lymphocytes also produce TNF-α. This is a pivotal cytokine that regulates an array of proinflammatory mediators. Recently, anti-TNF-α therapy using a chimeric anti-TNF-α monoclonal antibody (infliximab) and a TNF-receptor-immunoglobulin fusion protein (etanercept) have shown to be highly effective in patients with severe psoriasis. Efforts to treat psoriasis by inhibiting neovascularization of psoriatic plaques have also been shown to be effective. A randomized phase I/II clinical trial using Neovastat, a naturally occurring inhibitor of angiogenesis, resulted in dose-dependent improvement in the Psoriasis Area and Severity Index (PASI) score, thus providing further evidence that altered angiogenesis is an integral part of psoriasis pathophysiology. Since TM has proven antiangiogenic and anti-TNF-α activities, we are very encouraged that TM therapy will be beneficial in psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 + years of age
* Psoriasis vulgaris involving greater than 5% total body surface area
* No disease states or physical conditions which would impair evaluation of the test sites
* Willing and able to take test medications as directed in the protocol, make evaluation visits and follow protocol restrictions
* Failed systemic therapy for psoriasis (e.g., PUVA, retinoids, systemic steroids, methotrexate, etc.)
* Signed, written, witnessed informed consent form
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Use of any topical psoriasis treatment within weeks prior to the start of the study
* Use of any systemic medication within 4 weeks prior to the start of the study
* Involvement in an investigational study within the previous 4 weeks
* Inability to give informed consent
* History of drug dependency or alcoholism
* Severe infection within 4 weeks prior to study entry or the presence of chronic infection
* Significant psychiatric disorder
* Screening laboratory values which exceed the following limits:

  * Hematology - WBC <3,500 cells/mm3, Hb <10.5g/dl, platelets <100,000 cells/mm3;
  * Renal function test - creatinine >1.5 mg/dl;
  * Liver function tests - AST, alkaline phosphatase or total bilirubin more than twice the upper limits of normal, and a prothrombin time above the normal range.
* Pregnancy or breast feeding a baby. Sexually active women of reproductive age must use an acceptable form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Improvement in psoriasis as measured by PASI (psoriasis area and severity index)
Erythema, scaling, and thickness of target lesions

SECONDARY OUTCOMES:
Cytokine and laboratory values will be compared to baseline to test the hypothesis that TM will affect the level of TNF alpha, IL-1, C-protein, and TGF.

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States